CLINICAL TRIAL: NCT02639507
Title: International Consortium Investigating Early Vitrectomy in Diabetic Macular Edema Patients - the ICV-DME Study
Brief Title: International Consortium Investigating Early Vitrectomy in Diabetic Macular Edema Patients
Acronym: ICV-DME
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael W. Stewart, M.D., PI, Mayo Clinic
Other Study IDs: 14-008884
Record Dates: First submitted 2015-12-22; First posted 2015-12-24 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Diabetes With Diabetic Retinopathy With Macular Edema
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Vitrectomy

SUMMARY:
The purpose of this research is to evaluate the effectiveness of vitrectomy for the treatment of diabetic macular edema. Diabetes is known to cause retinal blood vessels to leak, leading to swelling of the central retina (macula), and decreased vision. Removing the vitreous gel with vitrectomy surgery is known to decrease the swelling caused by diabetes. Diabetic retinopathy is often treated with laser or injections of medicine in to the eye.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, > 18 years of age with type 1 or 2 diabetes mellitus diagnosed and treated by an endocrinologist, internist or family medicine physician
* Background diabetic retinopathy
* DME with central subfield thickness (CST) > 325 µm by Spectral Domain Optical Coherence Tomography (SD-OCT)
* HbA1c level of < 10.0 mg/dl
* Previous cataract surgery with implantation of a stable posterior chamber intraocular lens or a phakic eye with 1+ (out of 4+ scale) or less lens opacification
* Predominantly intact (80%) external limiting membrane (ELM) and photoreceptor inner/outer segment (IS/OS) lines within 500 µm of the fovea on horizontal and vertical SD-OCT scans
* Best corrected Snellen visual acuity from 20/40 to 20/280 inclusive.

Exclusion Criteria:

* Intraocular anti-vascular endothelial growth factor (VEGF) injection within the previous 3 months
* Systemic anti-VEGF or receptor tyrosine kinase inhibitor therapy within the previous 3 months
* Intraocular corticosteroid injection within the previous 6 months
* Peri-ocular corticosteroid injection within the previous 3 months
* Vitreomacular traction on SD-OCT scan (epiretinal membrane is allowed)
* Previous anterior or pars plana vitrectomy
* Glaucoma (IOP of > 21 mmHg or regular use of more than 2 IOP lowering drugs)
* Previous trabeculectomy
* Likelihood of needing intraocular surgery within 6 months
* Hard exudates involving the fovea
* Proliferative diabetic retinopathy with any evidence of retinal traction
* Cataract of grade 2+ or greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will have the following characteristics:
  * Background diabetic retinopathy.
  * Center involving macular edema with CST > 325 µm as measured by SD-OCT.
  * Predominantly intact (80%) ELM and IS/OS lines within 500 µm of the fovea on both horizontal and vertical SD-OCT scans.
  * Best corrected Snellen visual acuity from 20/40 to 20/280 inclusive
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
average (mean) improvement in Best Corrected Visual Acuity (BCVA) as measured with Snellen visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Stewart, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials